CLINICAL TRIAL: NCT00838032
Title: Pilot Study to Evaluate the Efficacy and Safety of Quetiapine Fumarate Instant-Release (Seroquel IR) in Controlling Agitation and Aggressive Symptoms in the Acute Treatment of Patients With Schizophrenia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Bo Zhang/ PhD., Mental Health Center of Huaxi Hospital affiliated to Sichuan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1443L00061
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2009-04-01 (Estimated); Status verified 2009-03

CONDITIONS: Acute Schizophrenia
Keywords: acute schizophrenic patients
MeSH Terms: interventions — Quetiapine Fumarate; Haloperidol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quetiapine fumarate (Experimental): Quetiapine fumarate should be initiated on Day 1 and titrated to at least 600 mg/day before Day 7 according to clinical experience and prescribe information. After Day 7, the dose of quetiapine fumarate should be adjusted between 600 mg/day to 750 mg/day at the discretion of the investigator.
  Interventions: Drug: Quetiapine fumarate
- Haloperidol (Active Comparator): Haloperidol should be initiated with the dose range from 5 mg/day to 15 mg/day from Day 1 to Day 5 (using injection) according to the clinical experience and prescribe information. After Day 7, the dose of haloperidol should be adjusted between 8 mg/day to 20 mg/day (change from injection to oral formulation between Day 6 to Day 7) at the discretion of the investigator.
  Interventions: Drug: Haloperidol

INTERVENTIONS:
Drug: Quetiapine fumarate — Quetiapine fumarate should be initiated on Day 1 and titrated to at least 600 mg/day before Day 7 according to clinical experience and prescribe information. After Day 7, the dose of quetiapine fumarate should be adjusted between 600 mg/day to 750 mg/day at the discretion of the investigator.
  Arms: Quetiapine fumarate
Drug: Haloperidol — Haloperidol should be initiated with the dose range from 5 mg/day to 15 mg/day from Day 1 to Day 5 (using injection) according to the clinical experience and prescribe information. After Day 7, the dose of haloperidol should be adjusted between 8 mg/day to 20 mg/day (change from injection to oral formulation between Day 6 to Day 7) at the discretion of the investigator.
  Arms: Haloperidol

SUMMARY:
Quetiapine fumarate is indicated for the treatment of patients with schizophrenia in China. Lots of clinical experience and evidence has demonstrated its efficacy and tolerability for the patient population. Some evidence showed that quetiapine fumarate could control aggression and agitation within 1 week, which is appropriate for the acute treatment of patients with schizophrenia. PANSS and MOAS are the common measurements for the efficacy of psychotic symptoms controlling in the clinical trials. Generally, 2 weeks are the appropriate timeframe for the evaluation of clinical effect of agitation and aggression symptoms controlling.

In adult patients with schizophrenia, quetiapine fumarate is licensed to maximal dose of 750mg/day. The target dose of quetiapine fumarate recommended in the manufacturer's prescribing information is 300-450 mg/day in China, though similar efficacy for quetiapine fumarate (600 mg/day), olanzapine (15 mg/day) and Risperidone (5 mg/day) was reported in a small, randomised, rater-blinded trial. Because of the low incidence of EPS, the limitation potential for weight gain and prolactin elevation, quetiapine fumarate should be well tolerated in this sensitive patient population with higher dose (600mg/day-750mg/day) (Peuskens 2004).

The aim of the present study is to evaluate the efficacy and safety of quetiapine fumarate with daily dose 600-750mg/day in improving agitation and aggression for the treatment of Chinese acute schizophrenic patients hospitalised for acute phase over a treatment period of 2 weeks

DETAILED DESCRIPTION:
Agitation and aggression are the common symptoms in the acute schizophrenic patients. Under these symptoms, schizophrenic patients could be harmful to themselves as well as the environment and people surrounding. Patients' agitation and aggression are also part of the reason for their hospitalisation. Therefore, rapid controlling of agitation and aggression for the patients is critical to ensure their treatment adherence, so that patients could stay with their treatment for a long time. Some studies have already provided the methods for rapid control, of which haloperidol is a common medication. However, use of haloperidol will bring patients prominent adverse reaction, such as extropyromidal symptoms etc., which will lead to the poor adherence of patients and caregivers and finally increase the treatment risk rather than benefit, such as relapse, re-hospitalization, and poor social functioning etc.

Quetiapine fumarate, a dibenzothiazepine derivative, is an atypical antipsychotic drug approved for treatment of schizophrenia, bipolar mania, and bipolar depression by FDA in many countries worldwide. In China, it has been used for the treatment of patients with schizophrenia for approximately 10 years. Quetiapine has the advantage of broad symptoms controlling, individualized dose range, and most important, good efficacy and tolerability in the acute treatment for schizophrenic patients.

Quetiapine fumarate is indicated for the treatment of patients with schizophrenia in China. Lots of clinical experience and evidence has demonstrated its efficacy and tolerability for the patient population. Some evidence showed that quetiapine fumarate could control aggression and agitation within 1 week, which is appropriate for the acute treatment of patients with schizophrenia. PANSS and MOAS are the common measurements for the efficacy of psychotic symptoms controlling in the clinical trials. Generally, 2 weeks are the appropriate timeframe for the evaluation of clinical effect of agitation and aggression symptoms controlling.

In adult patients with schizophrenia, quetiapine fumarate is licensed to maximal dose of 750mg/day. The target dose of quetiapine fumarate recommended in the manufacturer's prescribing information is 300-450 mg/day in China, though similar efficacy for quetiapine fumarate (600 mg/day), olanzapine (15 mg/day) and Risperidone (5 mg/day) was reported in a small, randomised, rater-blinded trial. Because of the low incidence of EPS, the limitation potential for weight gain and prolactin elevation, quetiapine fumarate should be well tolerated in this sensitive patient population with higher dose (600mg/day-750mg/day) (Peuskens 2004).

The aim of the present study is to evaluate the efficacy and safety of quetiapine fumarate with daily dose 600-750mg/day in improving agitation and aggression for the treatment of Chinese acute schizophrenic patients hospitalised for acute phase over a treatment period of 2 weeks This is a 2-week, single-blinded, randomised, parallel-group haloperidol-controlled pilot study. After given of informed consent and undergoing screening procedures, the patients will be allocated to study treatment on Day 1. Patients should have a diagnosis of schizophrenia by CCMD-3 criteria with MOAS total score at least 10. Eligible patients will be randomised into quetiapine group or haloperidol group with 1-week dose titration (at least 600 mg/day for quetiapine and 8 mg/day for haloperidol after Day 7). After that, the patients should be treated by the defined dose range for another week.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent by both patient and legal representative
2. A diagnosis of schizophrenia by Chinese Classification and Diagnostic Criteria of Mental Disorder, 3rd version (CCMD-3)
3. Male or female, aged 18 to 65 years
4. MOAS total score ³ 10 at both screening and randomization
5. Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at enrolment
6. Able to understand and comply with the requirements of the study

Exclusion Criteria:

1. Pregnancy or lactation
2. Any CCMD-3 not defined in the inclusion criteria
3. Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
4. Known intolerance or lack of response to quetiapine fumarate or haloperidol, as judged by the investigator
5. Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
6. Use of any of the following cytochrome P450 inducers in the 14 days preceding enrolment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
7. Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomisation
8. Substance or alcohol dependence at enrolment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by CCMD-3 criteria
9. Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by CCMD-3 criteria within 4 weeks prior to enrolment
10. Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
11. Unstable or inadequately treated medical illness (e.g. congestive heart failure, angina pectoris, hypertension) as judged by the investigator
12. Involvement in the planning and conduct of the study
13. Previous enrolment or randomisation of treatment in the present study.
14. Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements
15. A patient with Diabetes Mellitus (DM)
16. An absolute neutrophil count (ANC) of £ 1.5 x 109 per liter
17. 2 times higher than the normal upper limit of ALT or AST.
18. Use of clozapine within 28 days prior to randomisation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the efficacy of quetiapine fumarate in improving agitation and aggression symptoms for the schizophrenic patients | 14 days

SECONDARY OUTCOMES:
The response rate of quetiapine in improving agitation and aggression symptoms - the efficacy of quetiapine - the safety and tolerability of quetiapine - differences between quetiapine and haloperidol | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Tao Chun Liu, Director, Study Director — Huaxi hospital affiliated to Sichuan University
Locations (1):
- Mental Health Center of Huaxi Hospital affiliated to Sichuan University, Chengdu, Sichuan, China